CLINICAL TRIAL: NCT07149558
Title: Volume-Restricted Liver Resections for Perihilar Cholangiocarcinoma With Insufficient Future Liver Remnant Volume: A Prospective, Multicenter, Real-World Study
Brief Title: Volume-Restricted Resection for Perihilar Cholangiocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Yongjun Chen (Other)
Responsible Party: Sponsor-Investigator, Yongjun Chen, Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202507012
Record Dates: First submitted 2025-08-22; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cholangiocarcinoma, Hilar
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the safety and long-term outcomes of volume-restricted liver resection in patients with perihilar cholangiocarcinoma (pCCA) who have an insufficient future liver remnant (FLR). The main question it aims to answer is:

Does volume-restricted liver resection improve surgical safety and long-term survival compared with standard treatment in pCCA patients with insufficient FLR?

Participants with insufficient FLR who undergo volume-restricted liver resection or receive non-surgical treatment as part of their routine medical care will be followed for survival, postoperative complications, and other clinical outcomes. Data from patients with sufficient FLR undergoing standard radical resection will also be collected for comparison.

DETAILED DESCRIPTION:
Perihilar cholangiocarcinoma (pCCA) is a highly malignant tumor arising at the confluence of the right and left hepatic bile ducts. Its deep anatomical location and proximity to critical vascular structures render curative resection technically challenging and associated with substantial surgical risk. Surgical resection remains the only potentially curative treatment offering long-term survival. However, in some patients, an insufficient future liver remnant (FLR) precludes extensive hepatectomy, as it markedly increases the risk of postoperative liver failure and mortality, thereby limiting resectability and adversely affecting prognosis.

In recent years, volume-restricted liver resection has attracted growing interest. By ensuring negative bile duct margins while preserving as much functional liver parenchyma as possible, this approach may reduce the incidence of postoperative liver failure and improve both overall survival and quality of life. Nevertheless, prospective, multicenter, real-world evidence on the safety and efficacy of volume-restricted liver resection in pCCA patients with insufficient FLR remains scarce.

Against this background, the present study will target pCCA patients with insufficient FLR, implementing surgical strategies tailored to tumor extent and clinical presentation. These include perihilar resection, segment IVb resection, caudate-lobe-based resection (Taj Mahal procedure: resection of S1 + S4b + S5), and central hepatectomy (resection of S1 + S4 + S5 + S8). Outcomes will be compared with those of patients receiving non-surgical multimodal therapy, as well as with patients with sufficient FLR undergoing standard radical resection. By leveraging prospective, multicenter, real-world data, this study aims to evaluate the role of volume-restricted liver resection in improving surgical safety, reducing postoperative complications, and enhancing long-term survival, thereby providing evidence to refine surgical strategies for pCCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed hilar cholangiocarcinoma, or those with a high index of clinical suspicion for hilar bile duct malignancy despite the lack of histological confirmation.
* Patients who are able to understand and cooperate with this study.
* Patients who are able to provide and sign the written informed consent form before undergoing any screening procedures related to the study.

Exclusion Criteria:

* Patients with preoperatively or intraoperatively confirmed distant metastasis, including peritoneal dissemination, distant lymph node metastasis, hepatic or other organ metastasis.
* Patients who underwent palliative surgery only.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with perihilar cholangiocarcinoma and insufficient future liver remnant will be consecutively enrolled according to the inclusion and exclusion criteria. In addition, to better characterize the long-term survival of pCCA patients after surgical treatment, data from patients undergoing standard radical resection for pCCA will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of surgery/treatment until death or study termination, approximately 5 years.
  The period from the time when the patient was diagnosed with the disease or began receiving corresponding treatment until his or her death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival | Disease progression/death
  From the date the patient begins treatment to the date of disease progression or death, whichever occurs first.
R0 resection rate | Within 7 days after surgery(pathology report)
  The percentage of subjects achieving R0 resection.
90-day mortality | 90 days after the surgery
  The percentage of patients who died within 90 days among all patients.
Health-Related Quality of Life (HRQoL) | Surgical patients will receive monthly safety follow-ups (30 ± 7 days) for 3 months after discharge. All patients will have telephone survival/recurrence follow-ups every 2 months (60 ± 14 days) until death, loss to follow-up, or study end.
  HRQoL will be assessed during treatment follow-up using the EORTC QLQ-C30 questionnaire.
Incidence of postoperative complications | Within 90 days after the operation
  Defined as the percentage of patients who developed complications within 90 days after the operation among all included patients. Postoperative complications include bleeding, biliary fistula, abdominal cavity, liver failure, systemic inflammatory response syndrome (SIRS), gastrointestinal dysfunction, etc.